CLINICAL TRIAL: NCT00327301
Title: Systematic Characterization of the Cellular Proteome From Human Leukocytes of Glaucoma Patients in Comparison With Patients With Parkinson's Disease
Brief Title: Cellular Proteome From Leukocytes of Glaucoma Patients in Comparison With Patients With Parkinson's Disease
Status: Withdrawn | Type: Observational
Why Stopped: was replaced by an other study
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Bonn (Other)
Responsible Party: Sponsor
Other Study IDs: 075-WUK-2006-001
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Parkinson's Disease; Glaucoma
Keywords: POAG; Parkinson's disease; cellular proteome; human leucocytes; vasospasm; POAG patients; Patients with Parkinson's disease; Healthy subjects
MeSH Terms: conditions — Parkinson Disease; Glaucoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: None Retained — plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Glaucoma is a worldwide leading cause of blindness. The key feature of this ocular neuropathy is characterized by an excavating optic nerve head. Loss of retinal ganglion cells is the final end point in blinding diseases of the optic nerve such as glaucoma. It is known that neuronal cell death in glaucoma occurs by an apoptotic mechanism. In earlier studies the investigators could demonstrate that the process of apoptosis is reflected in circulating leukocytes by different parameters, like differential mRNA expression and an increased fragmentation of the DNA. Such alterations point out a relationship between cellular stress and apoptotic events.

Based on the results of mRNA-expression the investigators also expect alterations on the protein level.

This study is, therefore, designed to characterize the proteome related to the proteins involved in cell death related pathways.

Thus, the expression pattern of several proteins in leukocytes from patients with primary open angle glaucoma will be analyzed by techniques like Western-blot and tandem mass spectrometry. These samples will be compared with samples from healthy controls. In addition, they will also be compared with samples from patients with Parkinson's disease. Since glaucoma is a neurodegenerative disease, these patients will be included as positive controls in this study.

DETAILED DESCRIPTION:
Hypothesis:

Differences in the proteome concerning cell death pathways of glaucoma patients correspond to the differences in the mRNA expression of these patients.

Specific aims:

Characterization of the cellular proteome from human leukocytes of glaucoma patients compared to healthy controls and patients with Parkinson's disease.

Background:

Glaucoma is a worldwide leading cause of blindness. The key feature of this ocular neuropathy is characterized by an excavating optic nerve head. Loss of retinal ganglion cells is the final end point in blinding diseases of the optic nerve such as glaucoma. It is known that neuronal cell death in glaucoma occurs by an apoptotic mechanism. In earlier studies we could demonstrate that this cell death is reflected in circulating leukocytes by different parameters, like differential mRNA expression, and an increased fragmentation of the DNA. The differences in mRNA expression indicate a close relationship to cellular stress conditions and apoptotic events: increased mRNA expression was detected for p53, 20S proteasome alpha subunit, ABC1 transporter, p21(WAF1/CIP1), 14-3-3 sigma factor, MMP-9 and MMP-14, and TIMP-1.

Based on the assumption that glaucoma patients may differ on the level of their expression for these mRNAs, we expect that similar differences should exist at the protein level.

This study is, therefore, designed to characterize the proteome related to the proteins involved in cell death related pathways.

ELIGIBILITY:
Inclusion Criteria:

* German native speakers
* Age between 18-85 years
* Primary open-angle glaucoma (POAG) with and without vasospasm
* An inclusion criterion for one control group is Parkinson's disease.

Exclusion Criteria:

Any history of:

* Ocular or systemic diseases other than glaucoma or Parkinson's disease
* Drug or alcohol abuse
* Any condition potentially interfering with the visual field results. Visual fields will be obtained from the chart.
* Mental impairment interfering with the ability to cooperate and understand the purpose of this study; exception: those patients with Parkinson's disease. A prerequisite for including patients with Parkinson's disease in this study is the ability of these patients to cooperate and completely understand the purpose of this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: glaucoma patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Selim Orgül, MD, Study Director — University Hospital, Basel, Switzerland